CLINICAL TRIAL: NCT03751085
Title: A Clinical Study on Albert Wong Frame-based Stereotactic Biopsy System for Brain
Acronym: AWF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Lau Bik Liang, Dr., Ministry of Health, Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NMRR-17-3247-36799
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Intracranial CNS Disorder
Keywords: AW frame; biopsy; stereotactic; accuracy; safety
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AW frame (Experimental): AW frame biopsy
  Interventions: Device: AW frame

INTERVENTIONS:
Device: AW frame — AW stereotactic frame for intracranial lesion biopsy

SUMMARY:
This study is to establish a new, alternative stereotactic biopsy frame (AW frame) in the field of stereotactic neurosurgery.

DETAILED DESCRIPTION:
AW frame is a stereotactic biopsy frame created by Dr. Albert Sii Hieng Wong. A phantom study had completed by Dr. Bik Liang Lau and Dr. Albert Sii Hieng Wong in year 2017 with good accuracy. The phantom study result is going to be submitted for publication by early 2019.

With the good accuracy of AW frame in the phantom study, the frame has been approved by the Medical Research & ethic committee (MREC) for human use in a research setting.

In the study, patient with intracranial lesion which required biopsy, whom fulfilled the criteria will be recruited. All these patient will underwent standard biopsy procedure either under local or general anaesthesia with AW frame mounted.

A localisation CT scanning will be perform with localiser fixed onto the head frame. Target of the intracranial lesion is selected. The coordinates of the localizing points and the selected target inserted into the AW stereo-calculator to generate the AW frame setting up measurements.

Burr hole will be performed and biopsy taken by using Nashold® biopsy needle. An immediate post-biopsy CT imaging will be performed to confirm the site of the biopsy. Patient will be monitored in the neurosurgery ward for any complications.

Histopathologic analysis of the biopsies will be done using usual procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years old
* Radiological diagnosis of intracranial space occupying lesion of any etiology

Exclusion Criteria:

* Patient involved in other study trial
* Any serious medical condition that according to the investigator could interfere with the conduct of the study
* Unwillingness or inability to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-07-17 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | For each patient 2 week after the biopsy
  The diagnostic yield is defined as the number of patients in whom the histopathological diagnosis was made based of the biological material obtained during the biopsy.
Number of participants presenting with post-biopsy complications | an average of 2 week
  The presence of acute postoperative complication is noted if any of following findings is present: wound site infection up to two weeks after the biopsy, a new neurological deficit developed up to 24 hours following the operation and present in a follow up clinical examination 2 weeks postoperatively, intraparenchymal hematoma with radiological evidence.

SECONDARY OUTCOMES:
Time | From the time of the participant is transferred to the OR until the time of the participant transfer out of it, assessed on the day of operation.
  the preparation, operation and total operating room time
Length of hospital stay | an average of 1 week
  The preoperative, postoperative and total length of hospital stay

CONTACTS AND LOCATIONS:
Locations (3):
- Malaysia (3):
  - Department of Neurosurgery, Sarawak General Hospital, Kuching, Sarawak
  - Hospital Miri, Miri, Sarawak
  - Department of Neurosurgery, Hospital Sibu, Sibu, Sarawak

IPD SHARING:
Plan to Share IPD: No